CLINICAL TRIAL: NCT02669680
Title: Granulocyte Colony Stimulating Factor (G-CSF) to Treat Acute-on-chronic Liver Failure: A Multicentre Randomized Trial
Brief Title: Granulocyte Colony Stimulating Factor (G-CSF) to Treat Acute-on-chronic Liver Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Thomas Berg, Prof. Dr. med., University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRAFT
Record Dates: First submitted 2016-01-22; First posted 2016-02-01 (Estimated); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G-CSF + Standard therapy (Experimental): Standard care of acute-on-chronic liver failure and application of G-CSF
  Interventions: Drug: G-CSF; Other: Standard therapy
- Standard therapy (Active Comparator): Standard care of acute-on-chronic liver failure
  Interventions: Other: Standard therapy

INTERVENTIONS:
Drug: G-CSF — G-CSF subcutaneously, 5 μg/kg daily on day 0-4, then every 3rd day over 26 days (days 7, 10, 13, 16, 19, 22, 25) = 12 doses
  Other Names: Filgrastim
  Arms: G-CSF + Standard therapy
Other: Standard therapy

SUMMARY:
Multicentre, open, randomised, and controlled trial conducted in patients diagnosed with acute on chronic liver failure (ACLF) who meet inclusion/exclusion criteria.The objective of GRAFT-trial is to evaluate efficacy and safety of subcutaneously administered granulocyte colony-stimulating factor (G-CSF) in patients with ACLF. All patients will receive standard medical care for ACLF according to the guidelines. Patients in the experimental arm additional receive subcutaneous injections of G-CSF.

DETAILED DESCRIPTION:
The acute on chronic liver failure (ACLF) is characterised by a severe deterioration of liver function due to a precipitating event on top of an underlying chronic liver disease. As therapeutic options are limited the mortality rate lies between 40 and 80% at 3 months. The granulocyte colony-stimulating factor (G-CSF) mobilized stem- as well as immune cells and improved liver function in preclinical trials. G-CSF treatment reduced the rate of infectious complications and significantly improved patients´ survival in acute on chronic liver failure, shown recently in small randomised studies. Thus, G-CSF is a promising treatment option that needs to be evaluated in a multi-centre controlled trial. The GRAFT trial will randomise patients with ACLF between standard of care with and without G-CSF. All participants will be followed for 12 months in order to evaluate safety and efficacy of G-CSF. If successful, the GRAFT trial has the potential to change clinical practice in acute on chronic liver failure.

ELIGIBILITY:
Inclusion Criteria:

1. Acute-on-chronic liver failure (ACLF) according to the consensus criteria recently defined by the CANONIC study group [Moreau 2013]. Patients with acute decompensation of cirrhosis [defined as acute development of one or more of the following: ascites (onset and/or worsening), hepatic encephalopathy (onset and/or worsening), gastrointestinal haemorrhage, bacterial infection] are classified as ACLF if one of the following applies:

   * single kidney failure (serum creatinine level ≥ 2 mg/dl) or
   * single failure of one of the following organ systems: liver, coagulation, circulation, or respiration, together with a serum creatinine level ranging from 1.5 to < 2.0 mg/dl and/or mild to moderate hepatic encephalopathy or
   * single cerebral failure together with serum creatinine level ranging from 1.5 to < 2.0 mg/dl or
   * two or more organ failures. Organ failures are defined according to the CLIF-C OFs [Jalan 2014].
2. Age ≥ 18 years, male or female
3. Written informed consent from patient, legal or authorized representative or a confirmation of justification of trial participation by an independent medical consultant PLEASE NOTE: In case of confirmation by the independent medical consultant a deferred informed consent from patient, legal or authorized representative has to be given

Exclusion Criteria:

1. Prior not curatively treated or active malignancies
2. Sickle cell disease
3. septic shock, defined by the following symptom complex: bacteraemia AND SIRS AND shock
4. WBC-count of > 50 x 109/L
5. Known HIV infection
6. Known intolerance to filgrastim
7. Suspected lack of compliance
8. Pregnant or nursing women
9. Fertile women (within two years of their last menstruation) without appropriate contraceptive measures (implanon, injections, oral contraceptives, intrauterine devices, partner with vasectomy) while participating in the trial (participants using a hormone-based method have to be informed of possible effects from the trial medication on contraception).
10. Participation in other interventional trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Transplant-free survival up to 90 days (death or transplant count as events) | 90 days

SECONDARY OUTCOMES:
Overall survival time until the end of follow-up | 360 days
Transplant-free survival time until the end of follow-up | 360 days
Complications of ACLF (hepatorenal syndrome (HRS), variceal bleeding, ascites, hepatic encephalopathy (HE)) | 90 days/360 days
Infections (proven infection necessitating systemic use of antibiotics) | 90 days/360 days
Liver function - assessed by MELD-Score - during the course of treatment and follow-up | 360 days
Liver function - assessed by Child-Pugh-Score - during the course of treatment and follow-up | 360 days
Duration of the initial hospital stay | up to 360 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Berg, Prof., Study Director — University Hospital of Leipzig;
Locations (21):
- Germany (21):
  - University Hospital of Leipzig, Leipzig, Saxony
  - Universitätsklinikum Aachen, Aachen
  - Charité-Campus Virchow-Klinikum, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum KÖLN, Cologne
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Klinikum der J.W. Goethe- Universität, Frankfurt
  - Universitätsklinik Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Halle (Saale), Halle
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - HELIOS Park-Klinikum Leipzig, Leipzig
  - Klinikum St. Georg gGmbH, Leipzig
  - Universitätsklinikum Magdeburg AöR, Magdeburg
  - Universitätsmedizin Mainz, Mainz
  - Universitätsklinikum Tübingen, Tübingen
  - St. Josefs-Hospital, Wiesbaden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Engelmann C, Herber A, Franke A, Bruns T, Reuken P, Schiefke I, Zipprich A, Zeuzem S, Goeser T, Canbay A, Berg C, Trebicka J, Uschner FE, Chang J, Mueller T, Aehling N, Schmelzle M, Splith K, Lammert F, Lange CM, Sarrazin C, Trautwein C, Manns M, Haussinger D, Pfeiffenberger J, Galle PR, Schmiedeknecht A, Berg T. Granulocyte-colony stimulating factor (G-CSF) to treat acute-on-chronic liver failure: A multicenter randomized trial (GRAFT study). J Hepatol. 2021 Dec;75(6):1346-1354. doi: 10.1016/j.jhep.2021.07.033. Epub 2021 Aug 5. PMID 34364917
- See also: Link to the EU trials register to the GRAFT results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2015-002212-32/results

DOCUMENTS (1):
  • Study Protocol (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT02669680/Prot_000.pdf